CLINICAL TRIAL: NCT05617040
Title: A Phase 1/Phase 2 Trial to Evaluate Safety, Immunogenicity and PSA Response of VTP-850 Prostate Cancer Immunotherapeutic in Men With Biochemical Recurrence After Definitive Local Therapy for Prostate Cancer
Brief Title: Prime-boost Immunotherapeutic Trial in Men With Biochemical Recurrence After Definitive Local Therapy for Prostate Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The trial was discontinued following completion of the Phase 1 portion. This discontinuation was not based on safety concerns.
Sponsor: Barinthus Biotherapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PCA001
Record Dates: First submitted 2022-11-01; First posted 2022-11-15 (Actual); Results first posted 2025-11-10 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-10

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Phase 1 will follow a 3+3 design and determine the RP2R (dose level of both ChAdOx1-PCAQ and MVA-PCAQ, and route of administration of MVA-PCAQ) that will be used in Phase 2. Phase 2 will consist of 2 sequential stages. Stage 1 will enroll 19 additional participants at the RP2R. If 4 or more participants treated at the RP2R have a PSA response, Stage 2 will be opened to enrolment of up to 100 additional participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- IM/IM Low (Experimental): ChAdOx1-PCAQ 5*10^9 vp IM / MVA-PCAQ 5*10^7 pfu IM
  Interventions: Biological: ChAdOx1-PCAQ; Biological: MVA-PCAQ
- IM/IM Full (Experimental): ChAdOx1-PCAQ 2.5*10^10 vp IM / MVA-PCAQ 2*10^8 pfu IM
  Interventions: Biological: ChAdOx1-PCAQ; Biological: MVA-PCAQ
- IM/IV Full (Experimental): ChAdOx1-PCAQ 2.5*10^10 vp IM / MVA-PCAQ 2*10^7 pfu IV
  Interventions: Biological: ChAdOx1-PCAQ; Biological: MVA-PCAQ

INTERVENTIONS:
Biological: ChAdOx1-PCAQ — Recombinant nonreplicating chimpanzee adenovirus Oxford 1 (ChAdOx1) vector encoding 4 prostate cancer antigens: prostate-specific antigen (PSA), prostatic acid phosphatase (PAP), six-transmembrane epithelial antigen of prostate 1 (STEAP1), and an oncofoetal antigen (5T4).
Biological: MVA-PCAQ — Replication-deficient recombinant Modified Vaccinia virus Ankara (MVA) vector encoding the same prostate cancer antigens as ChAdOx1-PCAQ (prostate-specific antigen (PSA), prostatic acid phosphatase (PAP), six-transmembrane epithelial antigen of prostate 1 (STEAP1), and an oncofoetal antigen (5T4))

SUMMARY:
This is a multi-centre, Phase 1/2, open-label clinical trial of the VTP-850 prime-boost immunotherapeutic in men with biochemical recurrence after definitive local therapy for prostate cancer.

DETAILED DESCRIPTION:
This is a multi-center Phase 1/2 clinical trial to evaluate safety, PSA response, and immunogenicity of the VTP850 prime-boost immunotherapeutic in men with biochemical recurrence of prostate cancer (PCa) after definitive local therapy for PCa.

VTP-850 consists of 2 components: ChAdOx1-PCAQ and MVA-PCAQ. All participants will receive ChAdOx1-PCAQ on Day 1 (prime) and MVA-PCAQ on Days 29 and 57 (boosts; Intervention Period). Participants will be followed for 6 months or until start of new therapy such as Androgen Deprivation Therapy (ADT) or until development of unequivocal metastatic PCa (Short-term Follow-up Period). Participants who have a prostate-specific antigen (PSA) response, defined as ≥50% reduction in serum PSA compared to baseline at any time, measured twice consecutively, at least 2 weeks apart, during the 6 months follow up will be followed for an additional 18 months, up to 24 months from first dose, or until start of new therapy such as ADT or development of unequivocal metastatic PCa (Long-term Follow-up Period).

Phase 1 (15-18 participants) will follow a 3+3 design to determine the recommended phase 2 regimen (RP2R; dose level of both ChAdOx1-PCAQ and MVA-PCAQ, and route of administration of MVA-PCAQ (IM or IV)) that will be used in Phase 2.

Phase 2 will consist of 2 sequential stages. In Stage 1 of Phase 2, 19 additional participants will be enrolled at the chosen Phase 2 regimen. If 4 or more of the 25 participants at the RP2R (including the Phase 1 participants who received the same dose regimen) have a PSA response, Stage 2 will be opened to enrolment of up to 100 additional participants.

ELIGIBILITY:
Inclusion Criteria:

1. Males aged 18 years and above at the time of signing the informed consent.
2. Histologically or cytologically confirmed adenocarcinoma of the prostate.
3. Has undergone primary therapy for prostate cancer (radical prostatectomy and/or definitive external beam radiation and/or brachytherapy). Salvage external radiation therapy (XRT) following radical prostatectomy >6 months prior to Day 1 is allowed.
4. No further local therapy to prostate or systemic therapy for prostate cancer and no metastasis-directed therapy for PSA positron emission tomography (PET) positive lesions planned within 4 months after the first dose of VTP-850.
5. Serum testosterone >175 ng/dL.
6. Nonmetastatic (M0) disease and no evidence of prostatic bed recurrence verified by whole body bone scintigraphy and either CT or MRI. Note that a positive PSMA PET does not exclude the participant if the conventional scans are negative.
7. Serum PSA of >0.3 ng/mL for participants with prior radical prostatectomy (with or without salvage radiotherapy), or serum PSA of 2 ng/mL above nadir for participants with prior external beam radiation or brachytherapy.
8. PSA doubling time ≤12 months.
9. Not planning to start ADT for at least 4 months after Day 1.
10. Eastern Cooperative Oncology Group (ECOG) Score 0 or 1.
11. Baseline laboratory parameters must meet the following criteria:

    * Haemoglobin ≥110 g/L
    * White cell count ≥2.0×10^9/L
    * Absolute neutrophil count ≥1.5×10^9/L
    * Lymphocytes ≥0.9×10^9/L
    * Platelets ≥100×10^9/L
    * Creatinine ≤1.5×upper limit of normal (ULN) OR calculated creatinine clearance ≥50 mL/min by the Cockcroft Gault formula
    * Total bilirubin ≤1.5×ULN, (total bilirubin >1.5×ULN is acceptable if total bilirubin is fractionated and direct bilirubin <35%)
    * Alanine aminotransferase ≤1.5×ULN
    * Aspartate aminotransferase ≤1.5×ULN
    * Troponin T within normal range
    * HbA1c <7 %
12. Agrees to the following during the trial for at least 65 days after the last dose of VTP-850:

    * Refrain from donating sperm PLUS, either
    * Be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long-term and persistent basis) and agree to remain abstinent OR
    * Agrees to use a male condom when having sexual intercourse with a woman of childbearing potential, and should also be advised of the benefit for a female partner to use a highly effective method of contraception as a condom may break or leak.
13. Agrees to comply with all scheduled visits, VTP-850 administration plan, laboratory tests, lifestyle considerations and other trial procedures

Exclusion Criteria:

1. Any other prior malignancy within the past 5 years except for basal cell or squamous epithelial carcinomas of the skin that have been resected with no evidence of metastatic disease for 3 years.
2. Unstable medical condition, drug or alcohol abuse, or medical or psychiatric condition that in the opinion of the investigator would affect the safety of the participant or the evaluation of the data or interfere with adherence to the trial requirements.
3. Significant history of or current cardiovascular, respiratory, renal, gastrointestinal, endocrinological, haematological or neurological disorders constituting a risk when taking the trial intervention or interfering with the interpretation of data; cardiac event or heart failure in the previous 6 months.
4. Current or chronic history of liver disease. This includes but is not limited to: hepatitis virus infections, cirrhosis, drug- or alcohol-related liver disease, non alcoholic steatohepatitis, autoimmune hepatitis, hemochromatosis, Wilson's disease, α-1 antitrypsin deficiency, primary biliary cholangitis, primary sclerosing cholangitis or any other liver disease considered clinically significant by the investigator. (Note that history of hepatitis C infection, Gilbert's syndrome or non alcoholic fatty liver not associated with steatohepatitis are not exclusions. In line with Exclusion Criterion 10, active hepatitis C infection is exclusionary.)
5. Active autoimmune disease that has required systemic treatment in past 2 years with use of disease modifying agents, chronic corticosteroids (>14 days) or immunosuppressive drugs. Hormone replacement therapy (e.g., thyroxine, insulin or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is allowed.
6. History of severe allergy to eggs or history of severe reaction to any previous vaccination that required medical attention.
7. Medical history that could increase the participant's risk of reaction to a vaccine, including but not limited to capillary leak syndrome, transverse myelitis, multiple sclerosis, Guillain Barré syndrome, significant thrombocytopenia, thrombosis with thrombocytopenia syndrome (also termed vaccine-induced thrombotic thrombocytopenia), heparin-induced thrombocytopenia, or hereditary angioedema, acquired angioedema or idiopathic angioedema.
8. Any immunocompromised state, or history of solid organ or stem cell transplantation.
9. Active infection requiring parenteral antibiotic therapy or causing fever (temperature ≥38.0˚C) within 7 days prior to Day 1, or unexplained fever (temperature ≥38.0˚C) within 7 days prior to Day 1.
10. Known history of infection with hepatitis B virus, or human immunodeficiency virus, or active hepatitis C virus infection (antibody and RNA positive).
11. Received XRT following radical prostatectomy within 6 months prior to Day 1.
12. Received ADT outside of the initial primary therapy
13. Prior chemotherapy or immunotherapy (including vaccines or checkpoint inhibitors) or experimental agent or participation in a clinical trial for prostate cancer with the exception of those taking part as primary treatment option.
14. Received a vaccine with adenovirus vector within 3 months prior to Day 1.
15. Received any live vaccine within 30 days prior to Day 1, or planned vaccination to occur within 3 months after Day 1.
16. Received any non-live/inactivated vaccine within 14 days of Day 1 or planned non-live vaccination to occur within 10 weeks after Day 1.
17. Administration of immunoglobulins and/or any blood products within 28 days prior to Day 1.
18. Condition requiring systemic treatment with corticosteroids or other immunosuppressive medications within 14 days of first dose of VTP-850. Note that adrenal replacement doses are permitted. Inhaled and topical corticosteroids are allowed.
19. Received an investigational product or investigational surgical procedure in the 3 months prior to Day 1 or planned use during the trial period, or participation at any time in clinical trial for prostate cancer with exception of those taking part as primary treatment.
20. Any significant cardiovascular conditions per the investigator within 6 months before study entry including but not limited to: myocardial infarction, stroke, New York Heart Association class III or IV heart failure, thromboembolic events, major cardiovascular or cerebrovascular procedures, history of cardiac valvular disease or other structural heart disease or any other condition that in the investigator's opinion puts the participant at unacceptable risk to enter the study.
21. Participant with QT interval corrected for heart rate (QTc) determined using Fridericia's formula (QTcF; QTcF = QT/[R-R interval {RR}^0.33]) > 470 msec and any other ECG findings deemed clinically significant at screening.
22. Uncontrolled hypertension that, in the opinion of the Investigator, puts participant at increased risk of a cardiovascular event at the time of screening.
23. Uncontrolled dyslipidemia that, in the opinion of the Investigator, puts participant at increased risk of cardiovascular event at the time of screening.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male participants only
Enrollment: 22 (Actual)
Dates: Start 2023-01-30 (Actual); Primary Completion 2025-02-05 (Actual); Study Completion 2025-02-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Washington University School of Medicine, St Louis, Missouri
  - Columbia University Irving Medical Center, New York, New York
  - Cornell University, New York, New York
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - University of Virginia Health System, Charlottesville, Virginia
  - Fred Hutchinson Cancer Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | IM/IM Low | IM/IM Full | IM/IV Full
Started | 3 | 10 | 9
Completed | 3 | 9 | 8
Not Completed | 0 | 1 | 1
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Death | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IM/IM Low | IM/IM Full | IM/IV Full | Total
Number analyzed (Participants) | 3 | 10 | 9 | 22
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.0 (6.93) | 71.1 (4.89) | 68.9 (9.53) | 69.5 (7.25)
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 1 | 2
  White | 2 | 9 | 8 | 19
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 9 | 9 | 21
  Unknown or Not Reported | 0 | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 3 | 10 | 9 | 22

OUTCOME MEASURES:

1. Primary Outcome: The Safety of VTP-850 Prime-boost Regimens, With the Booster Dose Administered Either IM or IV, and the Recommended Phase 2 Regimen (RP2R)
Description: Participants with AEs, ≥Grade 3 AEs, and serious adverse events.
Time Frame: From the start of the first VTP-850 administration continuing until Month 6
Measure: Count of Participants; unit: Participants
Arm/Group | IM/IM Low | IM/IM Full | IM/IV Full
Number analyzed (Participants) | 3 | 10 | 9
Participants
  Participants with AEs | 3 | 9 | 9
  Grade 1 (Worst Severity) | 2 | 5 | 3
  Grade 2 (Worst Severity) | 1 | 4 | 5
  Grade 5 (Worst Severity) | 0 | 0 | 1
  Serious adverse events | 1 | 0 | 1

2. Secondary Outcome: The PSA Response Rate to VTP-850
Description: Percentage of participants with ≥50% reduction in serum PSA compared to baseline (2 consecutive measurements at least 2 weeks apart)
Time Frame: 6 months
Population: The Efficacy Evaluable Set (EES) will consist of all participants in the FAS who had one baseline measurement of PSA and at least one post-baseline measurement of PSA.
Measure: Count of Participants; unit: Participants
Arm/Group | IM/IM Low | IM/IM Full | IM/IV Full
Number analyzed (Participants) | 3 | 9 | 8
Participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From the start of the first VTP-850 administration continuing until Month 6
Arm/Group | IM/IM Low | IM/IM Full | IM/IV Full
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/10 | 1/9
Serious Adverse Events (participants affected / at risk) | 1/3 | 0/10 | 1/9
Other Adverse Events (participants affected / at risk) | 3/3 | 9/10 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IM/IM Low (N=3) | IM/IM Full (N=10) | IM/IV Full (N=9)
Death (General disorders) | 0 | 0 | 1
Cerebral ischaemia (Nervous system disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IM/IM Low (N=3) | IM/IM Full (N=10) | IM/IV Full (N=9)
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0
Fatigue (General disorders) | 0 | 3 | 3
Chills (General disorders) | 0 | 1 | 1
Injection site pain (General disorders) | 1 | 0 | 1
Injection site reaction (General disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 2 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 1
Irritability (Psychiatric disorders) | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Hot flush (Vascular disorders) | 1 | 1 | 0

LIMITATIONS AND CAVEATS:
The trial was initially designed as a Phase 1/2 trial; however, the sponsor elected to discontinue the trial following completion of the Phase 1 portion.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2024-04-18): https://cdn.clinicaltrials.gov/large-docs/40/NCT05617040/Prot_000.pdf
  • Statistical Analysis Plan (2024-10-31): https://cdn.clinicaltrials.gov/large-docs/40/NCT05617040/SAP_001.pdf